CLINICAL TRIAL: NCT07374484
Title: Longitudinal Dynamics of Angiotensin II Type 1 Receptor Antibodies Around Kidney Transplantation and Their Impact on Clinical Outcomes
Brief Title: Longitudinal Dynamics of AT1R Antibodies in Kidney Transplant Recipients
Acronym: AT1R
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Health, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Sang-Il Min, MD, PhD, Professor of Transplant Vascular Dapartment, Seoul National University Hospital
Other Study IDs: AT1R Antibodies in KT; RS-2023-KH140187 (Other Grant/Funding Number: Ministry of Health & Welfare, Republic of Korea)
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Kidney Transplantation; Graft Survival; Angiotensin II Type 1 Receptor Antibody
Keywords: Angiotensin II Type 1 Receptor Antibody; Kidney Transplantation; Graft Survival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the dynamics of Angiotensin II Type 1 Receptor Antibodies (AT1R-Ab) before and after kidney transplantation. The purpose is to understand how changes in AT1R-Ab levels may impact post-transplant kidney function and graft survival. Participants will include kidney transplant recipients, and their AT1R-Ab levels will be monitored over a one-year period. This research may help develop better predictive models for transplant outcomes, improving clinical decision-making for transplant physicians.

DETAILED DESCRIPTION:
The study will be conducted as a prospective cohort study involving kidney transplant recipients. The participants will undergo monitoring of their AT1R-Ab levels at multiple time points before and after the transplantation, including 2 weeks, 3 months, and 1 year post-transplant. Data collected will include clinical information such as kidney function tests, graft survival rates, and post-transplant complications. The study will aim to correlate AT1R-Ab dynamics with clinical outcomes such as delayed graft function (DGF), graft loss, and creatinine levels.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients were those who had serum samples collected at pre-transplant and at 2 weeks, 3 months, and 1-year post-transplant, with a minimum follow-up of 1 year

Exclusion Criteria:

Exclusion criteria were simultaneous multi-organ transplantation and age younger than 18 years.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was conducted at tertiary academic transplant center in South Korea and included kidney transplant recipients between 2016 and 2022. Eligible patients were those who had serum samples collected at pre-transplant and at 2 weeks, 3 months, and 1-year post-transplant, with a minimum follow-up of 1 year. Exclusion criteria were simultaneous multi-organ transplantation and age younger than 18 years. Among the 1,118 patients who underwent kidney transplantation during this period, 768 were excluded because they did not have at least four serum samples stored in the Seoul National University Hospital Biobank within 1 year after transplantation. Of the remaining 350 patients with four or more stored samples, 106 were excluded due to the absence of required time-point samples (pre-transplant and 2-week, 3-month, and 1-year post-transplant), and an additional 3 patients were excluded due to missing data for studied parameters. Consequently, a total of 241 patients were included.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Biopsy-Proven Acute Rejection (BPAR) within 3 years post-transplant | Up to 3 years post-transplant
  This study evaluates biopsy-proven acute rejection (BPAR) as the primary outcome, using protocol biopsies at 2 weeks and 1 year post-transplant.

SECONDARY OUTCOMES:
Renal Function: Serum Creatinine and eGFR at 2 weeks, 3 months, and 1 year post-transplant | At 2 weeks, 3 months, and 1 year post-transplant
  Secondary outcomes will include renal function, assessed by serum creatinine and eGFR at 2 weeks, 3 months, and 1 year post-transplant. The relationship between AT1R-Ab levels and renal function will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dragun D, Muller DN, Brasen JH, Fritsche L, Nieminen-Kelha M, Dechend R, Kintscher U, Rudolph B, Hoebeke J, Eckert D, Mazak I, Plehm R, Schonemann C, Unger T, Budde K, Neumayer HH, Luft FC, Wallukat G. Angiotensin II type 1-receptor activating antibodies in renal-allograft rejection. N Engl J Med. 2005 Feb 10;352(6):558-69. doi: 10.1056/NEJMoa035717. PMID 15703421
- [Background] Viboon S, Townamchai N, Phiancharoen S, Kupatawintu P, Dhitivat V, Nathalang O. Prevalence of Antibody against Angiotensin II Type 1 Receptor (AT1R) Among Thai Kidney Transplant Patients. Transplant Proc. 2018 Jun;50(5):1310-1315. doi: 10.1016/j.transproceed.2018.03.020. Epub 2018 Mar 12. PMID 29880351
- [Background] Kang ZY, Liu C, Liu W, Li DH. Effect of anti-angiotensin II type 1 receptor antibodies on the outcomes of kidney transplantation: a systematic review and meta-analysis. Nephrol Dial Transplant. 2022 May 25;37(6):1171-1180. doi: 10.1093/ndt/gfab344. PMID 34865146
- [Background] Sorohan BM, Ismail G, Leca N, Tacu D, Obrisca B, Constantinescu I, Baston C, Sinescu I. Angiotensin II type 1 receptor antibodies in kidney transplantation: An evidence-based comprehensive review. Transplant Rev (Orlando). 2020 Oct;34(4):100573. doi: 10.1016/j.trre.2020.100573. Epub 2020 Sep 25. PMID 33002671

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT07374484/Prot_SAP_000.pdf